CLINICAL TRIAL: NCT03784287
Title: A Multicenter, Multinational, Extension Study to Evaluate the Long Term Safety and Efficacy of Intracerebroventricular AX 250 in Patients With Mucopolysaccharidosis Type IIIB (MPS IIIB, Sanfilippo Syndrome Type B)
Brief Title: A Treatment Extension Study of Mucopolysaccharidosis Type IIIB
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Allievex Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AX 250-202
Record Dates: First submitted 2018-03-30; First posted 2018-12-21 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-10

CONDITIONS: Mucopolysaccharidosis Type IIIB; MPS III B
Keywords: Sanfilippo Syndrome Type B
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- AX 250 (Experimental): All subjects will receive AX 250 at the MTTD established in 250-201, 300mg administered weekly by ICV infusion that will continue for up to 240 weeks.
  Interventions: Drug: AX 250

INTERVENTIONS:
Drug: AX 250 — Chimeric fusion of recombinant human alpha-N-acetylglucosaminidase and truncated human insulin-like growth factor 2 (rhNAGLU-IGF2)

SUMMARY:
The primary objectives of this study are to evaluate the long-term safety and tolerability of AX 250 administered to subjects with MPS IIIB by an implanted ICV reservoir and catheter and to evaluate the impact of long-term AX 250 treatment on cognitive function in patients with MPS IIIB as assessed by developmental quotient (DQ).

ELIGIBILITY:
Inclusion Criteria:

* Must have completed 48 weeks in Part 2 of Study 250-201 and enter 250-202 within 8 weeks of study completion
* Written informed consent from parent or legal guardian and assent from subject, if required
* Has the ability to comply with protocol requirements, in the opinion of the investigator
* Males and females who are of reproductive age should practice true abstinence, defined as no sexual activity, during the study and for 6 months after the study has been completed (or withdrawal from the study). If sexually active and not practicing true abstinence, males and females of reproductive age must use a highly effective method of contraception while participating in the study.
* If female with childbearing potential, must have a negative pregnancy test at the Screening visit and be willing to have additional pregnancy tests during the study.

Exclusion Criteria:

* Has both (1) a cognitive AEq score ≤ 18 months, and (2) a DQ score ≤ 20
* Would not benefit from enrolling in the study in the opinion of the investigator
* Has received stem cell, gene therapy or ERT (other than AX 250) for MPS IIIB
* Has contraindications for neurosurgery (eg, congenital heart disease, severe respiratory impairment, or clotting abnormalities)
* Has contraindications for MRI scans (eg, cardiac pacemaker, metal fragment or chip in the eye, or aneurysm clip in the brain)
* Has a history of poorly controlled seizure disorder
* Is prone to complications from intraventricular drug administration, including patients with hydrocephalus or ventricular shunts
* Has received any investigational medication other than AX 250 within 30 days prior to the Baseline visit or is scheduled to receive any investigational drug during the course of the study
* Has a medical condition or extenuating circumstance that, in the opinion of the investigator, might compromise the subject's ability to comply with protocol requirements, the subject's well-being or safety, or the interpretability of the subject's clinical data.
* Is pregnant at any time during the study

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Evaluate the Long-term safety and tolerability of AX 250 administered in up to 33 subjects with MPS IIIB by assessing the number of participants with abnormal clinical laboratory values and/or Adverse Events related to the treatment | Entire study period, up to 240 weeks
Evaluating the impact of long-term AX 250 treatment on cognitive function in up to 33 patients with MPS IIIB as assessed by developmental quotient (DQ) | Entire study period, up to 240 weeks

SECONDARY OUTCOMES:
Evaluate the impact of long-term AX 250 treatment on cognitive function in up to 33 patients with MPS IIIB as assessed by age equivalent score (AEq) | Entire study period, up to 240 weeks
  Age equivalent score is derived from neurocognitive tests (Bayley Scales of Infant Development, 3rd edition OR Kaufman Assessment battery for Children, 2nd edition)
Characterize immunogenicity as measured by IgE levels, formation of anti-AX 250, IGF1 and IGF2 antibodies in Cerebrospinal fluid (CSF) and serum. | Entire study period, up to 240 weeks
Evaluate the impact of long-term AX 250 treatment on Heparan sulfate (HS) levels in cerebrospinal fluid (CSF), serum and urine. | Entire study period, up to 240 weeks
Evaluate the impact of long-term AX 250 treatment on brain structure assessed by magnetic resonance imaging (MRI) | Entire study period, up to 240 weeks
Evaluate the impact of long-term AX 250 treatment on adaptive function derived from the Vineland Adaptive Behavior Scales, 2nd edition (VABS-II) | Entire study period, up to 240 weeks
  VABS-II is a measure of adaptive behavior and can be used to assess the level of subjects' functioning at various ages. Scale ranges from 0-4 (0 meaning never performs the behavior, and 4 meaning almost always performs the behavior independently)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Allievex Corporation
Locations (8):
- United States (2):
  - Children's Hospital and Research Center Oakland, Oakland, California
  - UPMC Children's Hospital Pittburgh, Pittsburgh, Pennsylvania
- Fundación Cardio Infantil - Instituto de Cardiología, Bogotá, Colombia
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany
- Complexo Hospitalario Universitario de Santiago (CHUS) - Hospital Clínico Universitario, Santiago de Compostela, Spain
- MacKay Memorial Children's Hospital, Taipei, Taiwan
- Gazi University Faculty of Medicine, Ankara, Turkey (Türkiye)
- Great Ormond Street Hospital For Children, NHS Foundation Trust, London, United Kingdom